CLINICAL TRIAL: NCT02286388
Title: Multicenter Randomized Controlled Trial Comparing One-step Partial Caries Removal to Complete Caries Removal for the Treatment of Deep Carious Lesions in Permanent Teeth DECAT DEep CAries Treatment
Brief Title: Multicenter Trial Comparing One-step Partial Caries Removal to Complete Caries Removal for the Treatment of Deep Carious Lesions in Permanent Teeth. (DECAT : DEep CAries Treatment).
Acronym: DECAT
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-854
Record Dates: First submitted 2014-10-15; First posted 2014-11-07 (Estimated); Last update posted 2016-09-29 (Estimated); Status verified 2016-09

CONDITIONS: Deep Caries
Keywords: Deep carious lesion; incomplete caries removal; antibacterial adhesive system; dental composite resin; pulp vitality preservation; randomized controlled trial

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Partial excavation (Experimental): patients receiving after excavation (in case of absence of pulp exposure after excavation necessitating endodontic treatment) antibacterial adhesive or non-antibacterial adhesive
  Interventions: Procedure: A one-step partial caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Procedure: A complete caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Device: The application of an antibacterial dental adhesive (ClearfilTM SE Protect, Kuraray Dental).; Device: The application of a conventional dental adhesive (ClearfilTM SE Bond, Kuraray Dental)
- Complete excavation (Active Comparator): patients receiving after excavation (in case of absence of pulp exposure after excavation necessitating endodontic treatment) antibacterial adhesive or non-antibacterial adhesive
  Interventions: Procedure: A one-step partial caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Procedure: A complete caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Device: The application of an antibacterial dental adhesive (ClearfilTM SE Protect, Kuraray Dental).; Device: The application of a conventional dental adhesive (ClearfilTM SE Bond, Kuraray Dental)
- Antibacterial dental adhesive (Experimental): patients with prior partial or complete caries removal (excepted patients with a pulp exposure after excavation necessitating endodontic treatment)
  Interventions: Procedure: A one-step partial caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Procedure: A complete caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Device: The application of an antibacterial dental adhesive (ClearfilTM SE Protect, Kuraray Dental).; Device: The application of a conventional dental adhesive (ClearfilTM SE Bond, Kuraray Dental)
- Conventional dental adhesive (Active Comparator): patients with prior partial or complete caries removal (excepted patients with a pulp exposure after excavation necessitating endodontic treatment)
  Interventions: Procedure: A one-step partial caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Procedure: A complete caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth.; Device: The application of an antibacterial dental adhesive (ClearfilTM SE Protect, Kuraray Dental).; Device: The application of a conventional dental adhesive (ClearfilTM SE Bond, Kuraray Dental)

INTERVENTIONS:
Procedure: A one-step partial caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth. — Instruments and procedures:
  * Soprolife® (Acteon, La Ciotat, France) dental imaging device to detect dentinal infection status. The green-black light indicates infected dentin, red indicates infected/affected dentin and green indicates healthy dentinal tissue.
  * Sterile round bur under water spray coolant followed by final excavation with hand instruments The clinician will remove the superficial necrotic and demineralized dentin with complete excavation of the peripheral demineralized dentin, avoiding excavation close to the pulp.
  Hand instruments will be used for final excavation following clinical criteria guidelines (color of residual dentin and probe resistance) and taking in to consideration the color data obtained by the Soprolife® camera.
  The operator will stop excavating when the dentin close to the pulp appears red (for infected dentin).
Procedure: A complete caries removal procedure for the treatment of deep carious lesions in posterior permanent teeth. — Instruments and procedures:
  Idem partial excavation arm.
  In the complete excavation arm, the operator will stop excavating when the dentin close to the pulp appears green (for healthy dentin tissue) using the Soprolife® camera, leaving no infected or affected dentin.
Device: The application of an antibacterial dental adhesive (ClearfilTM SE Protect, Kuraray Dental). — Enamel and dentin will be conditioned according to the manufacturer's instructions. Both antibacterial and conventional adhesives are two-steps bonding systems.
  The first step consists of the application of a primer to the enamel and dentin for 20 seconds (which allows the completion of etching and priming procedures). The second step consists of the application of the antibacterial adhesive and its light curing for 10 seconds.
Device: The application of a conventional dental adhesive (ClearfilTM SE Bond, Kuraray Dental) — Idem antibacterial dental adhesive arm. A conventional dental adhesive will be used instead of an antibacterial.

SUMMARY:
This clinical trial is a national multicenter randomized controlled trial performed in parallel groups aiming to validate a treatment that preserves pulp vitality of mature permanent posterior teeth through partial removal of carious tissue and restoring tooth structure using a simple filling in one session, thus delaying premature tooth aging.

Two successive randomizations will be performed (allocation ratio 1:1); firstly for the type of excavation carried out (partial vs. complete caries removal) and secondly for the nature of the adhesive used (antibacterial adhesive vs. non-antibacterial adhesive). The second randomization will not be carried out for teeth requiring endodontic treatment after the first randomization.

The study's primary objective will be to compare, at 1 year of follow-up, the efficacy (binary success criteria) of partial caries removal versus complete caries removal in occlusal or proximal deep lesions of mature permanent posterior teeth (bicuspids and molars except third molars). Secondary objectives will include the comparison, at 1 year of follow-up, of the efficacy (binary success criteria) of an antibacterial two-step self-etch adhesive versus a traditional non-antibacterial two-step self-etch adhesive. Another secondary objective will be to compare, at two and three years of follow-up, the efficacy of partial versus complete caries removal.

The primary outcome is the success of the caries removal protocol at one year, measured according to 5 FDI criteria, while the secondary outcome is the contribution of the functional and biological dimensions of the 5 FDI criteria items to determining success or failure of the treatment. The outcome of success will be the same for all objectives, primary and secondary.

ELIGIBILITY:
Inclusion Criteria:

Randomization n°1 - Partial versus complete caries removal

Patient-related criteria:

* Patient consulting in one of the multicenter trial centers
* Male and female aged 8-80 (inclusive),
* Affiliated to a social security regimen
* Able to tolerate necessary restorative procedures
* Provide informed consent
* Accepts the three-year follow-up period

Tooth related criteria:

* Mature permanent posterior tooth
* Tooth with vital pulp according to pulp-sensitivity tests
* Tooth with a deep (primary or secondary) at least proximal and/or occlusal carious lesion presenting a residual dentin thickness with no continuity between the carious cavity and the pulp chamber.
* In case of proximal lesions, the proximal cervical limit must allow proper placement of a waterproof dental dam (confirmed by a bitewing X-ray radiograph)
* Tooth requiring a direct partial restorative treatment.

Randomization n°2 - Antibacterial vs. non antibacterial adhesive application

Tooth has been assigned a treatment by randomization n°1.

Exclusion Criteria:

Randomization n°1 - Partial versus complete caries removal

Patient-related criteria:

* Person under guardianship, pregnant or nursing woman,
* Risk of infectious endocarditis,
* Patient who has an implanted Cardiac Pacemaker/Defibrillator
* Patient with severe periodontal disease (pocket depth ≥5mm and/or mobility type IV),
* Poor oral hygiene (abundance of soft matter within the gingival pocket and/or on the tooth and gingival margin = score 3 [Silness and Loe, 1964],
* Allergy to any of the materials and/or anaesthetic used,
* Uncooperative patients.

Tooth related criteria:

* Nocturnal pain causing insomnia,
* Tooth suffering dentin hypersensitivity (sharp sudden pain of short duration pain arising from exposed dentin (erosion and/or gingival recession), typically in response to external stimuli (air blast hypersensitivity [Schiff et al., 1994], tactile hypersensitivity),
* Sensitivity to axial or lateral percussion;
* Radiolucent apical image,
* Condensing osteitis,
* Tooth having an external or internal resorption,
* Tooth having suffered trauma,
* Tooth with a carious cervical lesion,
* Tooth with an occlusal wear associated to a dentine exposure,
* Tooth supporting clasp of a removable partial denture (RPD).
* Tooth with defects of mineralization that once the treated tooth could come into contact of the carried out restoration

Randomization n°2 - Antibacterial vs. non antibacterial adhesive application

- Tooth with pulp exposure after randomization n°1 requiring endodontic treatment (pulp exposure > 2 mm² and/or haemostasis not obtained).

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 464 (Estimated)
Dates: Start 2015-02; Primary Completion 2017-08 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
Probability of success in arm P (Partial Caries Removal) compared to arm C (Complete Caries Removal) using a composite criteria of success summarized as a binary success criteria (cf. description below) | one year of follow-up.
  Cases will be considered as successful if each of the 5 following criteria described by the World Dental Federation (FDI) present a score of 3 or less:
  * Fracture of material and retention (item 5)
  * Marginal adaptation (item 6)
  * Radiographic examination (including apical pathologies) (item 9)
  * Post-operative sensitivity and tooth vitality (item 11)
  * Recurrence of caries (item 12) Criteria 5, 6 and 9 are functional criteria while criteria 11 and 12 are biological criteria.
  Considering a score of 4 or 5 as failure means that a re-intervention on the tooth (score 4) would be considered as a failure in the context of this study.
  Adverse events will be recorded and reported as general safety outcomes.

SECONDARY OUTCOMES:
Contribution of the functional and biological dimensions of the five FDI criteria items | At one year of follow-up.
  Assessment of the relative importance of each of the 5 FDI criteria in determining failure for both the primary outcome
Probability of success in arm P (Partial Caries Removal) compared to arm C (Complete Caries Removal) using a composite criteria of success summarized as a binary success criteria, at two and three years of follow-up. | At two and three years of follow-up.
  same criteria as the primary outcome measure of efficacy (composite criteria summarized as a binary success criteria)
Probability of success after the use of an antibacterial adhesive compared to the use of a non-antibacterial adhesive using a composite criteria of success summarized as a binary success criteria, at one, two and three years of follow-up. | At one, two and three years of follow-up.
  same criteria as the primary outcome measure of efficacy (composite criteria summarized as a binary success criteria)
Identification of predictive factors of clinical success from among the following list: presence of post-operative pain, age of patient, type of the carious lesion, location of the carious lesion (occlusal or proximal) and pulp exposure. | At one, two and three years of follow-up.
  the dependent variable (clinical success) corresponds to the same criteria as the primary outcome measure of efficacy (composite criteria summarized as a binary success criteria)
Description of the Consequences of Failures per Treatment Arm | At one, two and three years of follow-up.
  total number of visits, need for endodontic treatment, need for extraction

CONTACTS AND LOCATIONS:
Overall Officials: BRIGITTE GROSGOGEAT, Professor, Study Director — Hospices Civils de Lyon
Locations (15):
- France (15):
  - Hôpital Estaing, Clermont-Ferrand
  - Hôpital Albert Chenevier, Créteil
  - Cabinet Libéral, Grenay
  - Hôpital Charles Foix, Ivry-sur-Seine
  - CHU Lille, Lille
  - Service de consultations et traitements dentaires, Lyon
  - Hôpital de la Timone, Marseille
  - CHRU de Nantes, Nantes
  - CHU Nice, Nice
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Cabinet Libéral, Paris
  - APAH Rothschild- Garancière, Paris
  - Hopital Xavier Arnozan, Pessac
  - CHRU Rennes, Rennes
  - CHRU Toulouse, Toulouse

REFERENCES:
- [Derived] Villat C, Attal JP, Brulat N, Decup F, Domejean S, Dursun E, Fron-Chabouis H, Jacquot B, Muller Bolla M, Plasse-Pradelle N, Roche L, Maucort-Boulch D, Nony P, Gritsch K, Millet P, Gueyffier F, Grosgogeat B. One-step partial or complete caries removal and bonding with antibacterial or traditional self-etch adhesives: study protocol for a randomized controlled trial. Trials. 2016 Aug 15;17(1):404. doi: 10.1186/s13063-016-1484-0. PMID 27527342